CLINICAL TRIAL: NCT03184584
Title: An Open-Label Rollover Study of PBI 4050 in Subjects With Alström Syndrome
Brief Title: Open-Label Rollover Study of PBI 4050 in Subjects With Alström Syndrome
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated early due to redeployment of study site staff during Covid-19 pandemic
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-4050-CT-9-10
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Alström Syndrome
MeSH Terms: conditions — Alstrom Syndrome | interventions — setogepram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBI-4050 (Experimental)
  Interventions: Drug: PBI-4050

INTERVENTIONS:
Drug: PBI-4050 — Four 200 mg capsules (800 mg total) administered orally, once daily

SUMMARY:
Phase 2, open-label, single-arm, multi-centre study evaluating the long term safety and tolerability of PBI-4050 in subjects with Alström Syndrome who have completed a preceding ProMetic-sponsored Alström Syndrome study with PBI-4050.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, single-arm, multi-centre study evaluating the long term safety and tolerability of PBI-4050 in subjects with Alström Syndrome who have completed the end-of-treatment (EoT) visit in a preceding ProMetic-sponsored Alström Syndrome study with PBI-4050. This study will also evaluate the efficacy and pharmacological effects of PBI 4050 in this multi faceted disorder. Approximately 20 to 30 subjects will be enrolled to receive 800 mg PBI-4050 once daily for 96 weeks or until product licensing or study termination by the Sponsor, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed a preceding ProMetic-sponsored Alström syndrome study with PBI-4050.
* Subject has signed informed consent
* Subject has a documented diagnosis of Alström syndrome
* Subject receiving antidiabetic medications is able and willing to self-monitor blood glucose levels
* Subject must be willing to forego other forms of experimental drug treatment during the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening and agree to use adequate birth control from screening throughout the study and for 30 days after the last Investigational Medicinal Product (IMP) administration
* If a male subject has not been vasectomized at least 6 months before screening and partners with a woman of childbearing potential, he must be willing to use an acceptable contraceptive method throughout the study and for 30 days after the last IMP administration.

Exclusion Criteria:

* Subject discontinued PBI-4050 for safety reasons from any preceding ProMetic-sponsored Alström syndrome study with PBI-4050
* Subject has had a documented episode of severe hypoglycaemia within 12 months before screening and investigator judges that the subject is unable to adequately monitor their glucose levels.
* Subject has uncontrolled hypertension with BP > 170/100 mmHg as determined at screening.
* Woman who is pregnant, breast-feeding, or planning a pregnancy during the course of the study as determined at screening
* Subject has any condition that, in the investigator's opinion, is likely to interfere with study conduct and compliance
* Subject has a history of an allergic reaction to PBI-4050 or any of its excipients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal laboratory values and/or adverse events that are related to treatment | 96 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose over time | 96 weeks
Change from baseline in plasma insulin over time | 96 weeks
Change from baseline in glycated hemoglobin (HbA1c) over time | 96 weeks
Change from baseline in blood glucose as measured by weekly 4 point profile | 96 weeks
Change from baseline in the liver stiffness | 96 weeks
  Measured in kilopascal (kPa) correlated to fibrosis by using a FibroScan

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trus, Birmingham, United Kingdom